CLINICAL TRIAL: NCT02384707
Title: Reintroduction of Small Doses of Food in Allergic Children to Lightening the Elimination Diet.
Brief Title: Master Allergen Child Nutrition. Reintroduction of Small Doses
Acronym: MANOE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2010-A00448-31
Record Dates: First submitted 2014-11-24; First posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2014-11

CONDITIONS: Food Allergies
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- allergic food (Experimental): Reintroduction procedure for small doses :
  * Administration of the first dose the first dose must be allergic food or placebo
  * Clinical monitoring for 45 minutes
  * Administration of the second dose
  Interventions: Other: allegic food; Other: Placebo

INTERVENTIONS:
Other: allegic food — Reintroduction procedure for small doses :
  * Administration of the first dose
  * Clinical monitoring for 45 minutes
  * Administration of the second dose
Other: Placebo

SUMMARY:
Reintroduction of small doses of food in allergic children to lightening the elimination diet.

DETAILED DESCRIPTION:
In four groups of allergic children (peanuts, wheat , milk and egg), a reintroduction of 4 small increasing doses of allergen is carried out progressively double-blind placebo- cons , randomized, during a hospitalization.

The procedure for reintroduction of small doses (MPD) is stopped at the appearance of intolerance (in taking a dose of allergen or placebo) defined by the onset of allergic symptoms or objective severe abdominal pain within 45 minutes of taking.

ELIGIBILITY:
Inclusion Criteria:

* Allergic children 1 and 16 years for peanut, egg and wheat. So, for milk between 9 months and 16 years.
* Accurate diagnostic
* Allergic react rapidly and acute

Exclusion Criteria:

* severe disease

Ages: 9 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Tolerance for each ingested dose is assessed by a clinical score | 45 minutes
  Tolerance is defined by the absence of allergy symptoms within 45 minutes of ingestion of the allergen dose in the absence of intolerance to previous placebo

CONTACTS AND LOCATIONS:
Overall Officials: Martine Drouet, Principal Investigator — University Hospital, Angers
Locations (1):
- Denise Jolivot, Angers, Pays de Loire, France